CLINICAL TRIAL: NCT04417972
Title: A Phase I/II, Randomized, Double-Blind, Placebo-Controlled, Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics ,Pharmacodynamics and Efficacy of SHR7280 Tablets in Premenopausal Subjects With Endometriosis.
Brief Title: The Pharmacokinetic(PK)/Pharmacodynamics(PD) Study of SHR7280 Tablets in Premenopausal Subjects With Endometriosis.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR7280-102
Record Dates: First submitted 2020-05-21; First posted 2020-06-05 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- SHR7280 dose 1 (Experimental): oral administration for 21days,Phase I
  Interventions: Drug: SHR7280; Drug: Placebo oral tablet
- SHR7280 dose 2 (Experimental): oral administration for 21days,Phase I
  Interventions: Drug: SHR7280; Drug: Placebo oral tablet
- SHR7280 dose 3 (Experimental): oral administration for 21days,Phase I
  Interventions: Drug: SHR7280; Drug: Placebo oral tablet
- SHR7280 dose 4 (Experimental): oral administration for 21days,Phase I
  Interventions: Drug: SHR7280; Drug: Placebo oral tablet
- SHR7280 low dose (Active Comparator): oral administration for 84days,Phase II
  Interventions: Drug: SHR7280
- SHR7280 high dose (Active Comparator): oral administration for 84days, Phase II
  Interventions: Drug: SHR7280
- Placebo (Placebo Comparator): oral administration for 84days, Phase II
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: SHR7280 — treatment
  Arms: SHR7280 dose 1; SHR7280 dose 2; SHR7280 dose 3; SHR7280 dose 4; SHR7280 high dose; SHR7280 low dose
Drug: Placebo oral tablet — blank control
  Arms: Placebo; SHR7280 dose 1; SHR7280 dose 2; SHR7280 dose 3; SHR7280 dose 4

SUMMARY:
The primary objective of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of SHR7280 tablets in premenopausal subjects with endometriosis. In addition, this study will provide information on efficacy of SHR7280 tablets in premenopausal subjects with endometriosis.

DETAILED DESCRIPTION:
Endometriosis is a common disease, aﬀecting 5-10% of women of reproductive age . It is an estrogen-dependent and estrogen-driven disease and so hormonal manipulation and suppression of estrogen production form the basis of the majority of medical treatment. The primary objective of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of SHR7280 tablets in premenopausal subjects with endometriosis. In addition, this study will provide information on efficacy of SHR7280 tablets in premenopausal subjects with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

Phase I/II

1. premenopausal females, aged 18-45
2. History of regular menstrual cycles
3. Endometriosis participant diagnosed by surgical (e.g., laparoscopy or laparotomy) or by magnetic resonance imaging or ultrasonography.
4. Participant must agree to use only protocol specified rescue analgesics during the Screening and Treatment Periods for endometriosis-associated pain.
5. Participant in general good health. No clinically significant findings in laboratory parameters or clinically significant abnormality on X-ray Phase I (only) Participant has mild or moderate pelvic pain associated with endometriosis at Screening.

Phase II(only) Participant has moderate or severe pelvic pain associated with endometriosis at Screening.

Exclusion Criteria:

Phase I/II

1. Subjects with severe trauma or surgery within 6 months prior to the screening；
2. Known blood donation within 30 days pre-dose; donating≥200 ml of blood 2 months pre-dose;
3. Pregnant or Serum β-human chorionic gonadotropin (hCG)> 5 Million International Units(mIU)/mL at screening or baseline
4. Pregnant or breast feeding ;
5. Have pelvic pain that is not caused by endometriosis
6. Abnormal uterine bleeding
7. Are currently receiving gonadotropin-releasing hormone (GnRH) agonist, a GnRH antagonist or danazol or have received any of these agents within 6 months of the start of screening.
8. Are currently receiving subcutaneous medroxyprogesterone acetate (DMPA-SC) or intramuscular medroxyprogesterone acetate (DMPA-IM) or have received any of these agents within 3 months of the start of screening.
9. Are currently using hormonal contraception or other forms of hormonal therapy or received such treatment within 2 months of the start of screening.

Phase I (only) one month prior to screening involved in any drug or medical device clinical subjects, or within 5 half-life of drugs before screening; Phase II (only) Screening dual-energy x-ray absorptiometry (DXA) scan results of the lumbar spine, femoral neck, or total hip bone mineral density corresponding to 1.5 or more standard deviations below normal (T-score at or below -1.5)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 179 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse events | Pre-dose to 28±2 days after dose administration
  Phase I
Change From Baseline in the 7-day mean score for pelvic pain as measured by VAS at weeks 12 | Baseline and weeks 12
  Phase II daily assessment of dysmenorrhea score on a 4-point scale (0 = none, 1 = mild, 2 = moderate, 3 = severe) using an e-Diary.

SECONDARY OUTCOMES:
PK markers of SHR7280: area under the plasma concentration versus time curve (AUC) | At pre-defined intervals from initial dose through final study visit
  Phase I & II
PK markers of SHR7280: time to maximum plasma concentration(Tmax) | At pre-defined intervals from initial dose through final study visit
  Phase I & II
PK markers of SHR7280: maximum plasma concentration(Cmax) | At pre-defined intervals from initial dose through final study visit
  Phase I & II
PK markers of SHR7280: half-time(t1/2) | At pre-defined intervals from initial dose through final study visit
  Phase I & II
PK markers of SHR7280: apparent clearance(CL/F) | At pre-defined intervals from initial dose through final study visit
  Phase I & II
PK markers of SHR7280: apparent volume of distribution(Vz/F) | At pre-defined intervals from initial dose through final study visit
  Phase I & II
PD markers of SHR7280: Concentration of Estradiol(E2) | At pre-defined intervals from initial dose through final study visit
  Phase I & II
PD markers of SHR7280: Concentration of Progesterone(P) | At pre-defined intervals from initial dose through final study visit
  Phase I & II
PD markers of SHR7280: Concentration of Follicle stimulating hormone(FSH) | At pre-defined intervals from initial dose through final study visit
  Phase I & II
PD markers of SHR7280: Concentration of Luteinizing hormone(LH) | At pre-defined intervals from initial dose through final study visit
  Phase I & II
Change From Baseline in the 7-day mean score for pelvic pain as measured by VAS | Baseline and weeks 4、8
  Phase II
Change From Baseline in the Monthly Mean score for pelvic pain as measured by VAS | Baseline and weeks 4、8、12
  Phase II
Change From Baseline in the Monthly Mean Dysmenorrhea Score | Baseline and weeks 8、12
  Phase II
Change From Baseline in the Monthly Mean Non-menstrual Pelvic Pain Score and Dyspareunia Score | Baseline and weeks 4、8、12
  Phase II
Change from baseline to monthly analgesic use to treat endometriosis-associated pain | Baseline and weeks 4、8、12
  Phase II
Patient Global Impression of Change (PGIC) score at week 12 | Week 12
  Phase II
Adverse events | during Pre and 28±3 days after dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Hongyan Guo, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li Y, Zheng Y, Xu B, Cai L, Feng S, Liu Y, Zhu Z, Yu Q, Guo H. Safety, Pharmacokinetics, and Pharmacodynamics of SHR7280, a Non-peptide GnRH Antagonist in Premenopausal Women with Endometriosis: A Randomized, Double-Blind, Placebo-Controlled Phase 1 Study. Clin Pharmacokinet. 2023 Dec;62(12):1739-1748. doi: 10.1007/s40262-023-01315-6. Epub 2023 Oct 14. PMID 37838623